CLINICAL TRIAL: NCT03363594
Title: A Non-interventional Nationwide Registry to Identify Indian Phenotype Characteristics in Diabetes Mellitus Patients in India.
Brief Title: Indian Phenotype Registry
Acronym: IP Registry
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00282
Record Dates: First submitted 2017-11-20; First posted 2017-12-06 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes, T2D
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Diabetes Mellitus

SUMMARY:
This study is a non-interventional, multicentre observational study to be conducted at 1000 sites in India. The study targets to enrol approx. 50000 patients with approx. 50 patients per site. The study would enrol Diabetes Mellitus patients who provides written informed consent. No study medication will be prescribed or administered as a part of study procedure. Patients, who have been treated as per Investigators' routine clinical practice will be screened for enrolment in study. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB).

DETAILED DESCRIPTION:
This study is a non-interventional, multicentre observational study to be conducted at 1000 sites in India. The study targets to enrol approx. 50000 patients with approx. 50 patients per site. The study would enrol Diabetes Mellitus patients who provides written informed consent. No study medication will be prescribed or administered as a part of study procedure. Patients, who have been treated as per Investigators' routine clinical practice will be screened for enrolment in study. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB).

This is a single visit cross sectional study however during site feasibility visit, probability of follow-up of these patients will be evaluated. If feasible protocol will be amended to continue data collection prospectively for appropriate duration

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients with 18 years and above.
2. Patients who provide written informed consent.
3. Patients with previously diagnosed with Diabetes Mellitus
4. HbA1C report available within past 3 months

Exclusion Criteria- None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes Mellitus patients
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
To evaluate total body fat content across various BMI categories in the study population | 1 day
  Bioelectrical impedance will be used to estimate how much % body fat in terms of weight compared to total body weight.
  Since it is a ratio (weight of fat/total body weight) so no unit is required. The ratio will be multiplied by 100 to get Fat percentage.

SECONDARY OUTCOMES:
To analyse different characteristics of Diabetes Mellitus patient in study population | 1 day
  patient characteristics like age, gender
To correlate HbA1C level with various BMI categories | 1 day
  Weight in kilogram, height in meter will be combined to report BMI in kg/m2. then HbA1c in percentage and BMI in kg/m2 will be aggregated to get correlation

CONTACTS AND LOCATIONS:
Locations (197):
- India (197):
  - Research Site, Guntur, Andhra Pradesh
  - Research Site, Kākināda, Andhra Pradesh
  - Research Site, Madanapalle, Andhra Pradesh
  - Research Site, Nellore, Andhra Pradesh
  - Research Site, Rajahmundry, Andhra Pradesh
  - Research Site, Vijaywada, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Dibrugarh, Assam
  - Research Site, Guwahati, Assam
  - Research Site, Nagaon, Assam
  - Research Site, Silchar, Assam
  - Research Site, Tinsukia, Assam
  - Research Site, Bhagalpur, Bihar
  - Research Site, Gaya, Bihar
  - Research Site, Patna, Bihar
  - Research Site, Samāstipur, Bihar
  - Research Site, Samstipur, Bihar
  - Research Site, Bhilai, Chhattisgarh
  - Research Site, Durg, Chhattisgarh
  - Research Site, Raipur, Chhattisgarh
  - Research Site, Rohtak, Chhattisgarh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Amreli, Gujarat
  - Research Site, Anand, Gujarat
  - Research Site, Bharūch, Gujarat
  - Research Site, Bhavnagar, Gujarat
  - Research Site, Bhuj, Gujarat
  - Research Site, Borsad, Gujarat
  - Research Site, Botad, Gujarat
  - Research Site, Chaibasa, Gujarat
  - Research Site, Dohad, Gujarat
  - Research Site, Himatnagar, Gujarat
  - Research Site, Jamnagar, Gujarat
  - Research Site, Jūnāgadh, Gujarat
  - Research Site, Kutch, Gujarat
  - Research Site, Morvi, Gujarat
  - Research Site, Nadiād, Gujarat
  - Research Site, Navsari, Gujarat
  - Research Site, Pātan, Gujarat
  - Research Site, Porbandar, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Surat, Gujarat
  - Research Site, Unnao, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Valsād, Gujarat
  - Research Site, Vapi, Gujarat
  - Research Site, Bangalore, Haryana
  - Research Site, Faridabad, Haryana
  - Research Site, Gurugram, Haryana
  - Research Site, Hisar, Haryana
  - Research Site, Panchkula, Haryana
  - Research Site, Panipat, Haryana
  - Research Site, Rohtak, Haryana
  - Research Site, Sonīpat, Haryana
  - Research Site, Yamuna Nagar, Haryana
  - Research Site, Mandi, Himachal Pradesh
  - Research Site, Srinagar, Jammu and Kashmir
  - Research Site, Jamshedpur, Jharkhand
  - Research Site, Ranchi, Jharkhand
  - Research Site, Bangalore, Karnataka
  - Research Site, Belagavi, Karnataka
  - Research Site, Kalaburagi, Karnataka
  - Research Site, Angamaly, Kerala
  - Research Site, Chengannūr, Kerala
  - Research Site, Edappally, Kerala
  - Research Site, Ernākulam, Kerala
  - Research Site, Idukki, Kerala
  - Research Site, Kochi, Kerala
  - Research Site, Kollam, Kerala
  - Research Site, Kottayam, Kerala
  - Research Site, Malappuram, Kerala
  - Research Site, Nedumangād, Kerala
  - Research Site, Palakkad, Kerala
  - Research Site, Pezhakkappilly, Kerala
  - Research Site, Thalassery, Kerala
  - Research Site, Thiruvananthapuram, Kerala
  - Research Site, Thrissur, Kerala
  - Research Site, Trivandrum, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Guna, Madhya Pradesh
  - Research Site, Gwalior, Madhya Pradesh
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Jabalpur, Madhya Pradesh
  - Research Site, Mandsaur, Madhya Pradesh
  - Research Site, Ujjain, Madhya Pradesh
  - Research Site, Ahilyanagar, Maharashtra
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Bhiwandi, Maharashtra
  - Research Site, Kalyān, Maharashtra
  - Research Site, Kolhāpur, Maharashtra
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Navi Mumbai, Maharashtra
  - Research Site, Palanpur, Maharashtra
  - Research Site, Pālghar, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Raigad, Maharashtra
  - Research Site, Rajkot, Maharashtra
  - Research Site, Sangli, Maharashtra
  - Research Site, Satara, Maharashtra
  - Research Site, Sindhudurg, Maharashtra
  - Research Site, Solapur, Maharashtra
  - Research Site, Thane, Maharashtra
  - Research Site, Vasai, Maharashtra
  - Research Site, Imphal, Manipur
  - Research Site, Shillong, Meghālaya
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Berhampur, Odisha
  - Research Site, Bhubaneswar, Odisha
  - Research Site, Bhubneshwar, Odisha
  - Research Site, Bhuvaneshwar, Odisha
  - Research Site, Cuttack, Odisha
  - Research Site, Cuttuck, Odisha
  - Research Site, Paradip, Odisha
  - Research Site, Puri, Odisha
  - Research Site, Rourkela, Odisha
  - Research Site, Sambalpur, Odisha
  - Research Site, Amritsar, Punjab
  - Research Site, Jalandhar, Punjab
  - Research Site, Khanna, Punjab
  - Research Site, Kharar, Punjab
  - Research Site, Ludhiana, Punjab
  - Research Site, Moga, Punjab
  - Research Site, Patiāla, Punjab
  - Research Site, Ajmer, Rajasthan
  - Research Site, Ambala, Rajasthan
  - Research Site, Bikaner, Rajasthan
  - Research Site, Hanumāngarh, Rajasthan
  - Research Site, Jaipur, Rajasthan
  - Research Site, Jamshedpur, Rajasthan
  - Research Site, Jodhpur, Rajasthan
  - Research Site, Kota, Rajasthan
  - Research Site, Udaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Erode, Tamil Nadu
  - Research Site, Hosūr, Tamil Nadu
  - Research Site, Kanchipuram, Tamil Nadu
  - Research Site, Kochi, Tamil Nadu
  - Research Site, Kumbakonam, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Nagerkoil, Tamil Nadu
  - Research Site, Pattukkottai, Tamil Nadu
  - Research Site, Pondicherry, Tamil Nadu
  - Research Site, Ranipet, Tamil Nadu
  - Research Site, Salem, Tamil Nadu
  - Research Site, Thanjavur, Tamil Nadu
  - Research Site, Thiruvannamalai, Tamil Nadu
  - Research Site, Thiruvarur, Tamil Nadu
  - Research Site, Trichy, Tamil Nadu
  - Research Site, Vellore, Tamil Nadu
  - Research Site, Hyderabad, Telangana
  - Research Site, Karīmnagar, Telangana
  - Research Site, Secunderabad, Telangana
  - Research Site, Agra, Uttar Pradesh
  - Research Site, Aligarh, Uttar Pradesh
  - Research Site, Allahābād, Uttar Pradesh
  - Research Site, Bareilly, Uttar Pradesh
  - Research Site, Bareli, Uttar Pradesh
  - Research Site, Bulandshahr, Uttar Pradesh
  - Research Site, Etāwah, Uttar Pradesh
  - Research Site, Faizabad, Uttar Pradesh
  - Research Site, Firozabad, Uttar Pradesh
  - Research Site, Ghaziabad, Uttar Pradesh
  - Research Site, Gorakhpur, Uttar Pradesh
  - Research Site, Hāthras, Uttar Pradesh
  - Research Site, Jhānsi, Uttar Pradesh
  - Research Site, Kanpur, Uttar Pradesh
  - Research Site, Karnal, Uttar Pradesh
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Meerut, Uttar Pradesh
  - Research Site, Morādābād, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Piliphit, Uttar Pradesh
  - Research Site, Rāmpur, Uttar Pradesh
  - Research Site, Varanasi, Uttar Pradesh
  - Research Site, Dehradun, Uttarakhand
  - Research Site, Haldwani, Uttarakhand
  - Research Site, Baguihati, West Bengal
  - Research Site, Basīrhat, West Bengal
  - Research Site, Bolapur, West Bengal
  - Research Site, Burdwan, West Bengal
  - Research Site, Durgapur, West Bengal
  - Research Site, Guwahati, West Bengal
  - Research Site, Hābra, West Bengal
  - Research Site, Howrah, West Bengal
  - Research Site, Hubli, West Bengal
  - Research Site, Hugli, West Bengal
  - Research Site, Jalpāiguri, West Bengal
  - Research Site, Kharagpur, West Bengal
  - Research Site, Kolkata, West Bengal
  - Research Site, Malda, West Bengal
  - Research Site, Nabadwip, West Bengal
  - Research Site, Siliguri, West Bengal
  - Research Site, Chandigarh
  - Research Site, Goa

REFERENCES:
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00282&attachmentIdentifier=f06144e6-5b1b-4200-bd96-e4315aaf6d57&fileName=D1843R00282_CSR_synopsis_redacted.pdf&versionIdentifier=